CLINICAL TRIAL: NCT07210957
Title: The Effect of Manual Therapy in Individuals With Temporomandibular Disorders
Brief Title: Effect of Manual Therapy on Temporomandibular Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assoc. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-RK-12
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Temporomandibular Disorder; Neck Pain
Keywords: Ultrasound; Muscle Thickness; Manual Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Neck Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded, parallel, randomized controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Group allocation was concealed from participants, and outcome assessment was performed by a researcher who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy (Other): The manual therapy sessions implemented to individuals, will include one session per week for 6 weeks, will be lasted about 40-45 minutes. Myofascial techniques will be implemented to masseter, temporalis, suboccipital, scalene, levator scapula and trapezius muscles. These techniques will be lasted for 90 seconds and using with a sliding motion between the origin and insertion of the muscles. Dura mater (dural tube traction), suboccipital muscle release, pterygopalatine ganglion technique, and C0-C1-C2 mobilization as osteopathic techniques will be implemented.
  Interventions: Other: Manual Therapy
- Sham manual therapy (Sham Comparator): The control group will receive sham manual therapy protocol. Sham manual therapy includes implementations conducted under the same conditions and positions, however, without any therapeutic effect. The duration of each session will be lasted around 40-45 minutes (same as the therapy in the intervention group). The sham techniques will be implemented such as light contact by the therapist's hands, the impression of tissue manipulation, the touches with the effect of gravity and the performing non-therapeutic pressure to muscles.
  Interventions: Other: Sham manual therapy

INTERVENTIONS:
Other: Manual Therapy — Myofascial Release:
  Myofascial techniques will be implemented to masseter, temporalis, suboccipital, scalene, levator scapula and trapezius muscles. These techniques will be lasted for 90 seconds and using with a sliding motion between the origin and insertion of the muscles.
  Trigger Point Therapy:
  The ischemic compression approach will be implemented for 45-60 seconds to stretch the soft tissue over the trigger points of muscles. The emphasis will be on masseter, temporalis and scalene muscles
  . The emphasis will be on the fascial chains of cranio-cervical and cranio-mandibular transition areas.
  Arms: Manual therapy
Other: Sham manual therapy — The duration of each session will be lasted around 40-45 minutes (same as the therapy in the intervention group). The sham techniques will be implemented such as light contact by the therapist's hands, the impression of tissue manipulation, the touches with the effect of gravity and the performing non-therapeutic pressure to muscles. These sham techniques will not be implemented to the actual treatment points; however, they will be on the neck and jaw regions.
  Arms: Sham manual therapy

SUMMARY:
Temporomandibular disorders (TMD) are multifactorial conditions involving the temporomandibular joint and masticatory muscles, often presenting with pain and functional limitations. Conventional management includes splints, pharmacological approaches, physiotherapy, and manual therapy. This study aims to evaluate the effects of manual therapy compared to therapeutic exercise on muscle thickness, pain pressure threshold, range of motion, pain, mandibular function, and anxiety in individuals with TMD.

DETAILED DESCRIPTION:
TMD affects approximately one-quarter of the population and is characterized by pain, restricted movement, and impaired mandibular function. Etiology is multifactorial, including occlusal issues, trauma, bruxism, stress, and postural alterations. Bruxism in particular contributes to repetitive loading and hypertonia of the masticatory and cervical muscles, potentially influencing global posture. Current treatment approaches range from occlusal splints and surgery to conservative physiotherapy, manual therapy, and exercise. While manual therapy may reduce pain and restore mobility through techniques such as joint mobilization, myofascial release, and muscle inhibition, exercise supports improvements in strength, endurance, coordination, and joint stability. Evidence suggests that combined approaches may provide additive benefits. This trial will compare manual therapy and therapeutic exercise interventions in patients with TMD over six weeks. Objective outcomes will include ultrasound-based muscle thickness, pain pressure threshold, mandibular range of motion, pain intensity, and mandibular function. Anxiety levels will also be assessed using validated questionnaires. The primary hypothesis is that manual therapy will produce greater improvements across these measures compared to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Myalgia, and both myalgia and arthralgia according to Diagnostic Criteria for Temporomandibular Disorders
* Completing signing the informed consent form

Exclusion Criteria:

* Any rheumatological or metabolic disease
* Receiving any treatment for temporomandibular joint in the last 2 years (such as botulinum toxin, manual therapy, splint, orthodontics)
* A history of traumatic temporomandibular joint
* A history of diagnosed psychological diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Ultrasound Assessment | Baseline, sixth week
  Muscle thickness of the masseter and temporalis will be measured with a linear probe in neutral rest and during submaximal teeth clenching (supine). The probe will be aligned to standard anatomical landmarks, kept perpendicular to the skin without compressing soft tissue. Thickness will be recorded in millimeters as the distance between the internal and external fascia. Each muscle will be assessed once per condition.

SECONDARY OUTCOMES:
Pain Pressure Threshold | Baseline, sixth week
  A handheld algometer (1 cm² probe tip, 0-40 kg/cm² range, 0.1 kg increments) will be applied perpendicularly to the masseter, temporalis, upper trapezius, suboccipital muscles, and the C5 facet joint bilaterally. Participants will signal at first pain. Three measurements per site will be taken at 30-second intervals; the mean value (kg/cm²) will be used.
Maximum Mouth Opening and Lateral Excursion | Baseline, sixth week
  Measured in millimeters using a manual ruler between the upper and lower central incisors. Maximum unassisted opening will be recorded in supine. For lateral excursion, participants will move the mandible to the right and left as far as possible; distances will be recorded for each side. Pain or discomfort will be noted.
Mandibular Function Scale | Baseline, sixth week
  Self-report questionnaire with two parts: functional activities (speaking, smiling, chewing, etc.) and nutrition (difficulty with oral feeding). Each item is scored 0 (no difficulty) to 4 (severe difficulty). Higher total scores indicate greater dysfunction.
State-Trait Anxiety Inventory | Baseline, sixth week
  Consists of 40 items: 20 assessing state anxiety and 20 assessing trait anxiety. Each item is scored 1-4, giving subscale totals of 20-80. Higher scores indicate higher anxiety.
Generalized Anxiety Disorder Scale | Baseline, sixth week
  A 7-item self-report questionnaire assessing generalized anxiety over the past 2 weeks. Each item is scored 0 (not at all) to 3 (nearly every day). Total score ranges 0-21; scores 5, 10, and 15 represent cut-offs for mild, moderate, and severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: numan yener, phd, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University Department of Physiotherapy and Rehabilitation, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The dataset can be obtained from the principal investigator upon any reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: After publication
Access Criteria: via mail ramazankurul@ibu.edu.tr